CLINICAL TRIAL: NCT02878161
Title: Screening Protein Predictive of Response to Tumor Necrosis Factor-α Inhibitors Treatment in Chinese Rheumatoid Arthritis From "Real World" and Investigating Its Mechanism Through Signal Pathway
Brief Title: Predictability Studies on the Efficacy of TNF-α Inhibitors in Chinese RA From "Real World"
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fen Li (Other)
Responsible Party: Sponsor-Investigator, Fen Li, associate chief physician, Central South University
Organization: Central South University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: XYEYY-GZ81571599-20160118-1
Record Dates: First submitted 2016-07-12; First posted 2016-08-25 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; tumor necrosis factor α inhibitor; predictive; iTRAQ; signal pathway
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab; Etanercept; Adalimumab; Leflunomide; Licensure; Anti-Inflammatory Agents, Non-Steroidal; Glucocorticoids; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A group (Experimental): Infliximab plus Methotrexate , Leflunomide and NSAIDs and Glucocorticoids are permitted but not necessary included.
  Interventions: Drug: methotrexate(necessary); Biological: infliximab; Drug: leflunomide (permitted, not necessary); Drug: NSAIDs (permitted,not necessary); Drug: Glucocorticoids (permitted,not necessary)
- B group (Experimental): Etanercept plus Methotrexate , Leflunomide and NSAIDs and Glucocorticoids are permitted but not necessary included.
  Interventions: Drug: methotrexate(necessary); Biological: etanercept; Drug: leflunomide (permitted, not necessary); Drug: NSAIDs (permitted,not necessary); Drug: Glucocorticoids (permitted,not necessary)
- C group (Experimental): Adalimumab plus Methotrexate , Leflunomide and NSAIDs and Glucocorticoids are permitted but not necessary included.
  Interventions: Drug: methotrexate(necessary); Biological: adalimumab; Drug: leflunomide (permitted, not necessary); Drug: NSAIDs (permitted,not necessary); Drug: Glucocorticoids (permitted,not necessary)

INTERVENTIONS:
Drug: methotrexate(necessary) — Methotrexate will be received orally with dosage of 10mg/ week for every patient and MTX dose must be stable for at least 4 weeks.
  Other Names: MTX
Biological: infliximab — infliximab :intravenous injection 200mg,every times,0,2,6,14week ,4 times)
  Other Names: IFX
  Arms: A group
Biological: etanercept — Etanercept :hypodermic injection,25mg/twice a week
  Other Names: ETN
  Arms: B group
Biological: adalimumab — Adalimumab:hypodermic injection,40mg/twice a week
  Other Names: ADA
  Arms: C group
Drug: leflunomide (permitted, not necessary) — LEF will be permitted if patient had received for 1 month before enrollment and will not be changed for 14 weeks.
  Other Names: LEF
Drug: NSAIDs (permitted,not necessary) — NSAIDs will be allowed if patient had received for 1 month before enrollment and will not be changed for 14 weeks.
  Other Names: non steroidal anti inflammatory drugs
Drug: Glucocorticoids (permitted,not necessary) — Glucocorticoids (prednisone less than 10mg/day, or equal dosage of other similar drugs) will be permitted if the patient had received for 1 month before enrollment and the dosage will not be changed during the period.
  Other Names: prednisone,methylprednisolone,etc.

SUMMARY:
Rheumatoid arthritis (RA) is a chronic and disabling disease. tumor necrosis factor-a(TNF-a) inhibitors have demonstrated an outstanding performance in relieving joint inflammation and retarding bone erosion involved in RA. However, there is still about one-thirds of RA patients had a poor response to TNF α inhibitors. The Investigators hope to discover prediction protein with a domestic genetic background and finally establish prediction system with Chinese characteristics.

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a chronic and disabling disease. TNF-α inhibitors have demonstrated an outstanding performance in relieving joint inflammation and retarding bone erosion involved in RA. However, there is still about one-thirds of RA patients had a poor response to TNF α inhibitors. Currently the personalized biological treatment is the research hotspot. Recent studies focuses on exploring biomarkers predictive of drug response. The research methods such as genomics, transcriptomics, proteomics, metabolomics and immunocytology, have been applied,but they are not successfully integrated. The related studies in China are still at an initial stage, which necessitates an in-depth study in this area. The investigators' preliminary study showed that TNF-α-308 gene polymorphisms existed in Chinese RA patients and phosphoinositide 3-kinase/Akt signal pathway was activated in proliferated synovial fibroblasts stimulated by TNF-α. Therefore, for the first attempt in China, the investigators intend to screen for differential proteins by using isobaric tags for relative and absolute quantitation(iTRAQ) technique in RA patients receiving anti-TNF-α therapy, and then verify the predictive effects of selected differential proteins from the upstream gene polymorphism to the downstream protein expression. The investigators will also explore the mechanisms of differential proteins involved in TNF-α related signal pathway by using in vitro gene transfer, siRNA interference, and RA animal models. Through this study investigator hope to discover some prediction proteins with a domestic genetic background and finally establish a prediction system with Chinese characteristics.

ELIGIBILITY:
Inclusion Criteria:

* signed the consents voluntarily
* age between 18-75 years old
* patients were meet the American College of Rheumatology(ACR)

  * European League Against Rheumatism(EULAR) 2009 diagnostic criteria (total scores beyond 6)
* for severe RA patients DAS28-CRP≥5.1
* The participants receiving Infliximab plus Methotrexate will be invited to enroll the study.
* The participants receiving Etanercept plus Methotrexate will be invited to enroll the study.
* The participants receiving Adalimumab plus Methotrexate will be invited to enroll the study.

Exclusion Criteria:

* The patient have the disease history or the disease of cardiovascular, respiratory system, liver, gastrointestinal tract, endocrine, hematology, neurology or psychiatric disturbance, and investigator believe that there are some risks for patients with these disease history or disease when use study drugs, or these disease history or disease will disturb the interpret of data
* Patients with cancer in situ or exist the possibility of cancer malignancies
* Basically or completely loss of mobility, lack self-care ability, such as rely on a wheelchair or bed-ridden .
* Experimental examination display any of the following:

Aspartate aminotransferase or alanine aminotransferase>1.5 times of the upper limit of the normal value Total bilirubin>1.5 times of the upper limit of the normal value Total white blood cells <2500 cells/L absolute neutrophil count <1200 cells/L lymphocyte count <750 cells/L platelet<100000/L

* Patients with symptomatic herpes simplex
* Latent tuberculosis signal (PPD+++ OR T-SPOT>5 )
* Positive result of the hepatitis B virus (HBV):

HBsAg + Or HBeAg + Or HBeAg + Or HBcAb + Or HBV DNA +

* hepatitis C virus(HCV)+ or HCV RNA +
* HIV infection or HIV+
* 1 months before join the group, from a clinical point of view,patients have a serious infection caused by the virus, bacteria, fungi, or parasites
* Pregnancy 、 location 、prepare for conceive in one years or there is risk to impregnate their partners
* Patients received any biological therapies for 6 months, or participated any other clinical trials of new drugs
* A history of drug allergy
* A history of heavy drink
* vaccinate the live vaccine recently

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
EULAR (European League Against Rheumatism) response will be assessed among patients of 3 groups | Baseline, Weeks 14
  EULAR (European League Against Rheumatism) response is based on changes of DAS28-CRP. The following good, moderate and no response are defined based on changes of DAS28-CRP from baseline to weeks 14: >1.2 units are good response; 0.6-1.2 units are moderate response; ≤0.6 units are no response.
  The DAS28-CRP will be calculated at every visit within the clinical database. The components of the DAS28-CRP score assessment are: Tender/Painful Joint Count (28); Swollen Joint Count (28), hsCRP, and the Subject General Health VAS assessment. This efficacy measurement will be made at baseline and weeks 14.

SECONDARY OUTCOMES:
The changes of TNF level with different EULAR response will be assessed among patients of 3 groups. | Baseline, Weeks 14
  The TNF level assessment is a direct measurement using ELISA by testing patients' serum. This measurement will be made at baseline and weeks 14.
  The classification of EULAR response and the calculation of DAS28-CRP are based on above of Primary Outcome Measure.
The changes of Interest proteins with different EULAR response will be assessed among patients of 3 group. | Baseline, Weeks 14
  Interest proteins will be screened by iTRAQ (isobaric tags for relative and absolute quantitation). This measurement will be made at baseline and weeks 14 by comparing part of patients with good response or no response.
  Interest proteins being screened will be verified by Western Blot among all patients of 3 groups.
  The classification of EULAR response and the calculation of DAS28-CRP are based on above of Primary Outcome Measure.
The SNP (Single nucleotide polymorphism) of gene about TNF with different EULAR response will be assessed among patients of 3 groups. | Weeks 14
  SNP of TNF gene will be tested by PCR-RFLP (Polymerase Chain Reaction -Restriction Fragment Length Polymorphism). This measurement will be made at weeks 14 among all 3 groups' patients.
  The classification of EULAR response and the calculation of DAS28-CRP are based on above of Primary Outcome Measure.
The SNP of gene about interest proteins with different EULAR response will be assessed among patients of 3 groups. | Weeks 14
  SNP of gene about interest proteins will tested by PCR-HRM(Polymerase Chain Reaction-high resolution melting). This measurement will be made at weeks 14 among all 3 groups' patients.
  Interest proteins are screened and verified on above of Secondary Outcome Measure.
  The classification of EULAR response and the calculation of DAS28-CRP are based on above of Primary Outcome Measure.

CONTACTS AND LOCATIONS:
Overall Officials: Fen Li, doctor, Principal Investigator — Second Xiangya Hospital of Central South University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Vollenhoven RF. Switching between anti-tumour necrosis factors: trying to get a handle on a complex issue. Ann Rheum Dis. 2007 Jul;66(7):849-51. doi: 10.1136/ard.2007.069872. PMID 17576784
- [Background] Radstake TR, Svenson M, Eijsbouts AM, van den Hoogen FH, Enevold C, van Riel PL, Bendtzen K. Formation of antibodies against infliximab and adalimumab strongly correlates with functional drug levels and clinical responses in rheumatoid arthritis. Ann Rheum Dis. 2009 Nov;68(11):1739-45. doi: 10.1136/ard.2008.092833. Epub 2008 Nov 19. PMID 19019895
- [Background] Miossec P, Verweij CL, Klareskog L, Pitzalis C, Barton A, Lekkerkerker F, Reiter S, Laslop A, Breedveld F, Abadie E, Flamion B, Dere W, Mpofu S, Goel N, Ethgen D, Mitlak B, Ormarsdottir S, Rao R, Tsouderos Y, Reginster JY; Group for Respect of Ethics and Excellence in Science (GREES). Biomarkers and personalised medicine in rheumatoid arthritis: a proposal for interactions between academia, industry and regulatory bodies. Ann Rheum Dis. 2011 Oct;70(10):1713-8. doi: 10.1136/ard.2011.154252. Epub 2011 Jul 22. PMID 21784723
- [Background] Zeng Z, Duan Z, Zhang T, Wang S, Li G, Gao J, Ye D, Xu S, Xu J, Zhang L, Pan F. Association between tumor necrosis factor-alpha (TNF-alpha) promoter -308 G/A and response to TNF-alpha blockers in rheumatoid arthritis: a meta-analysis. Mod Rheumatol. 2013 May;23(3):489-95. doi: 10.1007/s10165-012-0699-5. Epub 2012 Jul 4. PMID 22760475
- [Background] Kang CP, Lee KW, Yoo DH, Kang C, Bae SC. The influence of a polymorphism at position -857 of the tumour necrosis factor alpha gene on clinical response to etanercept therapy in rheumatoid arthritis. Rheumatology (Oxford). 2005 Apr;44(4):547-52. doi: 10.1093/rheumatology/keh550. Epub 2005 Feb 3. PMID 15695296
- [Background] Miceli-Richard C, Comets E, Verstuyft C, Tamouza R, Loiseau P, Ravaud P, Kupper H, Becquemont L, Charron D, Mariette X. A single tumour necrosis factor haplotype influences the response to adalimumab in rheumatoid arthritis. Ann Rheum Dis. 2008 Apr;67(4):478-84. doi: 10.1136/ard.2007.074104. Epub 2007 Aug 2. PMID 17673491
- [Background] Nishimoto T, Seta N, Anan R, Yamamoto T, Kaneko Y, Takeuchi T, Kuwana M. A single nucleotide polymorphism of TRAF1 predicts the clinical response to anti-TNF treatment in Japanese patients with rheumatoid arthritis. Clin Exp Rheumatol. 2014 Mar-Apr;32(2):211-7. Epub 2013 Dec 9. PMID 24321457
- [Background] Potter C, Hyrich KL, Tracey A, Lunt M, Plant D, Symmons DP, Thomson W, Worthington J, Emery P, Morgan AW, Wilson AG, Isaacs J, Barton A; BRAGGSS. Association of rheumatoid factor and anti-cyclic citrullinated peptide positivity, but not carriage of shared epitope or PTPN22 susceptibility variants, with anti-tumour necrosis factor response in rheumatoid arthritis. Ann Rheum Dis. 2009 Jan;68(1):69-74. doi: 10.1136/ard.2007.084715. Epub 2008 Mar 28. PMID 18375541
- [Background] Padyukov L, Lampa J, Heimburger M, Ernestam S, Cederholm T, Lundkvist I, Andersson P, Hermansson Y, Harju A, Klareskog L, Bratt J. Genetic markers for the efficacy of tumour necrosis factor blocking therapy in rheumatoid arthritis. Ann Rheum Dis. 2003 Jun;62(6):526-9. doi: 10.1136/ard.62.6.526. PMID 12759288
- [Background] Davila-Fajardo CL, Marquez A, Pascual-Salcedo D, Moreno Ramos MJ, Garcia-Portales R, Magro C, Alegre-Sancho JJ, Balsa A, Cabeza-Barrera J, Raya E, Martin J. Confirmation of -174G/C interleukin-6 gene promoter polymorphism as a genetic marker predicting antitumor necrosis factor treatment outcome. Pharmacogenet Genomics. 2014 Jan;24(1):1-5. doi: 10.1097/FPC.0000000000000013. PMID 24253594
- [Background] Coulthard LR, Taylor JC, Eyre S; Biologics in Rheumatoid Arthritis Genetics and Genomics; Robinson JI, Wilson AG, Isaacs JD, Hyrich K, Emery P, Barton A, Barrett JH, Morgan AW, McDermott MF. Genetic variants within the MAP kinase signalling network and anti-TNF treatment response in rheumatoid arthritis patients. Ann Rheum Dis. 2011 Jan;70(1):98-103. doi: 10.1136/ard.2010.133249. Epub 2010 Aug 30. PMID 20805296
- [Background] Potter C, Cordell HJ, Barton A, Daly AK, Hyrich KL, Mann DA, Morgan AW, Wilson AG; Biologics in Rheumatoid Arthritis Genetics and Genomics Study Syndicate (BRAGGSS); Isaacs JD. Association between anti-tumour necrosis factor treatment response and genetic variants within the TLR and NFkappaB signalling pathways. Ann Rheum Dis. 2010 Jul;69(7):1315-20. doi: 10.1136/ard.2009.117309. Epub 2010 May 6. PMID 20448286
- [Background] Tan RJ, Gibbons LJ, Potter C, Hyrich KL, Morgan AW, Wilson AG, Isaacs JD; BRAGGSS; Barton A. Investigation of rheumatoid arthritis susceptibility genes identifies association of AFF3 and CD226 variants with response to anti-tumour necrosis factor treatment. Ann Rheum Dis. 2010 Jun;69(6):1029-35. doi: 10.1136/ard.2009.118406. Epub 2010 May 5. PMID 20444755
- [Background] Cui J, Saevarsdottir S, Thomson B, Padyukov L, van der Helm-van Mil AH, Nititham J, Hughes LB, de Vries N, Raychaudhuri S, Alfredsson L, Askling J, Wedren S, Ding B, Guiducci C, Wolbink GJ, Crusius JB, van der Horst-Bruinsma IE, Herenius M, Weinblatt ME, Shadick NA, Worthington J, Batliwalla F, Kern M, Morgan AW, Wilson AG, Isaacs JD, Hyrich K, Seldin MF, Moreland LW, Behrens TW, Allaart CF, Criswell LA, Huizinga TW, Tak PP, Bridges SL Jr, Toes RE, Barton A, Klareskog L, Gregersen PK, Karlson EW, Plenge RM. Rheumatoid arthritis risk allele PTPRC is also associated with response to anti-tumor necrosis factor alpha therapy. Arthritis Rheum. 2010 Jul;62(7):1849-61. doi: 10.1002/art.27457. PMID 20309874
- [Background] Krintel SB, Essioux L, Wool A, Johansen JS, Schreiber E, Zekharya T, Akiva P, Ostergaard M, Hetland ML. CD6 and syntaxin binding protein 6 variants and response to tumor necrosis factor alpha inhibitors in Danish patients with rheumatoid arthritis. PLoS One. 2012;7(6):e38539. doi: 10.1371/journal.pone.0038539. Epub 2012 Jun 7. PMID 22685579
- [Background] Liu C, Batliwalla F, Li W, Lee A, Roubenoff R, Beckman E, Khalili H, Damle A, Kern M, Furie R, Dupuis J, Plenge RM, Coenen MJ, Behrens TW, Carulli JP, Gregersen PK. Genome-wide association scan identifies candidate polymorphisms associated with differential response to anti-TNF treatment in rheumatoid arthritis. Mol Med. 2008 Sep-Oct;14(9-10):575-81. doi: 10.2119/2008-00056.Liu. PMID 18615156
- [Background] Cui J, Stahl EA, Saevarsdottir S, Miceli C, Diogo D, Trynka G, Raj T, Mirkov MU, Canhao H, Ikari K, Terao C, Okada Y, Wedren S, Askling J, Yamanaka H, Momohara S, Taniguchi A, Ohmura K, Matsuda F, Mimori T, Gupta N, Kuchroo M, Morgan AW, Isaacs JD, Wilson AG, Hyrich KL, Herenius M, Doorenspleet ME, Tak PP, Crusius JB, van der Horst-Bruinsma IE, Wolbink GJ, van Riel PL, van de Laar M, Guchelaar HJ, Shadick NA, Allaart CF, Huizinga TW, Toes RE, Kimberly RP, Bridges SL Jr, Criswell LA, Moreland LW, Fonseca JE, de Vries N, Stranger BE, De Jager PL, Raychaudhuri S, Weinblatt ME, Gregersen PK, Mariette X, Barton A, Padyukov L, Coenen MJ, Karlson EW, Plenge RM. Genome-wide association study and gene expression analysis identifies CD84 as a predictor of response to etanercept therapy in rheumatoid arthritis. PLoS Genet. 2013 Mar;9(3):e1003394. doi: 10.1371/journal.pgen.1003394. Epub 2013 Mar 28. PMID 23555300
- [Background] Umicevic Mirkov M, Cui J, Vermeulen SH, Stahl EA, Toonen EJ, Makkinje RR, Lee AT, Huizinga TW, Allaart R, Barton A, Mariette X, Miceli CR, Criswell LA, Tak PP, de Vries N, Saevarsdottir S, Padyukov L, Bridges SL, van Schaardenburg DJ, Jansen TL, Dutmer EA, van de Laar MA, Barrera P, Radstake TR, van Riel PL, Scheffer H, Franke B, Brunner HG, Plenge RM, Gregersen PK, Guchelaar HJ, Coenen MJ. Genome-wide association analysis of anti-TNF drug response in patients with rheumatoid arthritis. Ann Rheum Dis. 2013 Aug;72(8):1375-81. doi: 10.1136/annrheumdis-2012-202405. Epub 2012 Dec 11. PMID 23233654
- [Background] Marquez A, Ferreiro-Iglesias A, Davila-Fajardo CL, Montes A, Pascual-Salcedo D, Perez-Pampin E, Moreno-Ramos MJ, Garcia-Portales R, Navarro F, Moreira V, Magro C, Caliz R, Ferrer MA, Alegre-Sancho JJ, Joven B, Carreira P, Balsa A, Vasilopoulos Y, Sarafidou T, Cabeza-Barrera J, Narvaez J, Raya E, Canete JD, Fernandez-Nebro A, Ordonez Mdel C, de la Serna AR, Magallares B, Gomez-Reino JJ, Gonzalez A, Martin J. Lack of validation of genetic variants associated with anti-tumor necrosis factor therapy response in rheumatoid arthritis: a genome-wide association study replication and meta-analysis. Arthritis Res Ther. 2014 Mar 11;16(2):R66. doi: 10.1186/ar4504. PMID 24612463
- [Background] Lindberg J, Wijbrandts CA, van Baarsen LG, Nader G, Klareskog L, Catrina A, Thurlings R, Vervoordeldonk M, Lundeberg J, Tak PP. The gene expression profile in the synovium as a predictor of the clinical response to infliximab treatment in rheumatoid arthritis. PLoS One. 2010 Jun 25;5(6):e11310. doi: 10.1371/journal.pone.0011310. PMID 20593016
- [Background] Pachot A, Arnaud B, Marrote H, Cazalis MA, Diasparra J, Gouraud A, Mougin B, Miossec P. Increased tumor necrosis factor-alpha mRNA expression in whole blood from patients with rheumatoid arthritis: reduction after infliximab treatment does not predict response. J Rheumatol. 2007 Nov;34(11):2158-61. Epub 2007 Sep 15. PMID 17896807
- [Background] Sekiguchi N, Kawauchi S, Furuya T, Inaba N, Matsuda K, Ando S, Ogasawara M, Aburatani H, Kameda H, Amano K, Abe T, Ito S, Takeuchi T. Messenger ribonucleic acid expression profile in peripheral blood cells from RA patients following treatment with an anti-TNF-alpha monoclonal antibody, infliximab. Rheumatology (Oxford). 2008 Jun;47(6):780-8. doi: 10.1093/rheumatology/ken083. Epub 2008 Apr 3. PMID 18388148
- [Background] Julia A, Erra A, Palacio C, Tomas C, Sans X, Barcelo P, Marsal S. An eight-gene blood expression profile predicts the response to infliximab in rheumatoid arthritis. PLoS One. 2009 Oct 22;4(10):e7556. doi: 10.1371/journal.pone.0007556. PMID 19847310
- [Background] Stuhlmuller B, Haupl T, Hernandez MM, Grutzkau A, Kuban RJ, Tandon N, Voss JW, Salfeld J, Kinne RW, Burmester GR. CD11c as a transcriptional biomarker to predict response to anti-TNF monotherapy with adalimumab in patients with rheumatoid arthritis. Clin Pharmacol Ther. 2010 Mar;87(3):311-21. doi: 10.1038/clpt.2009.244. Epub 2009 Dec 23. PMID 20032971
- [Background] Meugnier E, Coury F, Tebib J, Ferraro-Peyret C, Rome S, Bienvenu J, Vidal H, Sibilia J, Fabien N. Gene expression profiling in peripheral blood cells of patients with rheumatoid arthritis in response to anti-TNF-alpha treatments. Physiol Genomics. 2011 Apr 12;43(7):365-71. doi: 10.1152/physiolgenomics.00127.2010. Epub 2011 Jan 25. PMID 21266503
- [Background] Wright HL, Thomas HB, Moots RJ, Edwards SW. Interferon gene expression signature in rheumatoid arthritis neutrophils correlates with a good response to TNFi therapy. Rheumatology (Oxford). 2015 Jan;54(1):188-93. doi: 10.1093/rheumatology/keu299. Epub 2014 Aug 13. PMID 25125592
- [Background] Fabre S, Dupuy AM, Dossat N, Guisset C, Cohen JD, Cristol JP, Daures JP, Jorgensen C. Protein biochip array technology for cytokine profiling predicts etanercept responsiveness in rheumatoid arthritis. Clin Exp Immunol. 2008 Aug;153(2):188-95. doi: 10.1111/j.1365-2249.2008.03691.x. Epub 2008 Jun 18. PMID 18549443
- [Background] Hueber W, Tomooka BH, Batliwalla F, Li W, Monach PA, Tibshirani RJ, Van Vollenhoven RF, Lampa J, Saito K, Tanaka Y, Genovese MC, Klareskog L, Gregersen PK, Robinson WH. Blood autoantibody and cytokine profiles predict response to anti-tumor necrosis factor therapy in rheumatoid arthritis. Arthritis Res Ther. 2009;11(3):R76. doi: 10.1186/ar2706. Epub 2009 May 21. PMID 19460157
- [Background] Trocme C, Marotte H, Baillet A, Pallot-Prades B, Garin J, Grange L, Miossec P, Tebib J, Berger F, Nissen MJ, Juvin R, Morel F, Gaudin P. Apolipoprotein A-I and platelet factor 4 are biomarkers for infliximab response in rheumatoid arthritis. Ann Rheum Dis. 2009 Aug;68(8):1328-33. doi: 10.1136/ard.2008.093153. Epub 2008 Jul 29. PMID 18664547
- [Background] Visvanathan S, Rahman MU, Keystone E, Genovese M, Klareskog L, Hsia E, Mack M, Buchanan J, Elashoff M, Wagner C. Association of serum markers with improvement in clinical response measures after treatment with golimumab in patients with active rheumatoid arthritis despite receiving methotrexate: results from the GO-FORWARD study. Arthritis Res Ther. 2010;12(6):R211. doi: 10.1186/ar3188. Epub 2010 Nov 17. PMID 21083889
- [Background] Sakthiswary R, Shaharir SS, Mohd Said MS, Asrul AW, Shahril NS. IgA rheumatoid factor as a serological predictor of poor response to tumour necrosis factor alpha inhibitors in rheumatoid arthritis. Int J Rheum Dis. 2014 Nov;17(8):872-7. doi: 10.1111/1756-185X.12443. Epub 2014 Oct 7. PMID 25292482
- [Background] Mathsson L, Mullazehi M, Wick MC, Sjoberg O, van Vollenhoven R, Klareskog L, Ronnelid J. Antibodies against citrullinated vimentin in rheumatoid arthritis: higher sensitivity and extended prognostic value concerning future radiographic progression as compared with antibodies against cyclic citrullinated peptides. Arthritis Rheum. 2008 Jan;58(1):36-45. doi: 10.1002/art.23188. PMID 18163519
- [Background] Morozzi G, Fabbroni M, Bellisai F, Cucini S, Simpatico A, Galeazzi M. Low serum level of COMP, a cartilage turnover marker, predicts rapid and high ACR70 response to adalimumab therapy in rheumatoid arthritis. Clin Rheumatol. 2007 Aug;26(8):1335-8. doi: 10.1007/s10067-006-0520-y. Epub 2007 Feb 7. PMID 17285224
- [Background] Gonzalez-Alvaro I, Ortiz AM, Tomero EG, Balsa A, Orte J, Laffon A, Garcia-Vicuna R. Baseline serum RANKL levels may serve to predict remission in rheumatoid arthritis patients treated with TNF antagonists. Ann Rheum Dis. 2007 Dec;66(12):1675-8. doi: 10.1136/ard.2007.071910. Epub 2007 Jul 31. PMID 17666448
- [Background] Mavragani CP, La DT, Stohl W, Crow MK. Association of the response to tumor necrosis factor antagonists with plasma type I interferon activity and interferon-beta/alpha ratios in rheumatoid arthritis patients: a post hoc analysis of a predominantly Hispanic cohort. Arthritis Rheum. 2010 Feb;62(2):392-401. doi: 10.1002/art.27226. PMID 20112385
- [Background] Choi IY, Gerlag DM, Herenius MJ, Thurlings RM, Wijbrandts CA, Foell D, Vogl T, Roth J, Tak PP, Holzinger D. MRP8/14 serum levels as a strong predictor of response to biological treatments in patients with rheumatoid arthritis. Ann Rheum Dis. 2015 Mar;74(3):499-505. doi: 10.1136/annrheumdis-2013-203923. Epub 2013 Dec 2. PMID 24297376
- [Background] Kapoor SR, Filer A, Fitzpatrick MA, Fisher BA, Taylor PC, Buckley CD, McInnes IB, Raza K, Young SP. Metabolic profiling predicts response to anti-tumor necrosis factor alpha therapy in patients with rheumatoid arthritis. Arthritis Rheum. 2013 Jun;65(6):1448-56. doi: 10.1002/art.37921. PMID 23460124
- [Background] Chen DY, Chen YM, Chen HH, Hsieh CW, Lin CC, Lan JL. Increasing levels of circulating Th17 cells and interleukin-17 in rheumatoid arthritis patients with an inadequate response to anti-TNF-alpha therapy. Arthritis Res Ther. 2011 Jul 30;13(4):R126. doi: 10.1186/ar3431. PMID 21801431
- [Background] Ceeraz S, Hall C, Choy EH, Spencer J, Corrigall VM. Defective CD8+CD28+ regulatory T cell suppressor function in rheumatoid arthritis is restored by tumour necrosis factor inhibitor therapy. Clin Exp Immunol. 2013 Oct;174(1):18-26. doi: 10.1111/cei.12161. PMID 23786396
- [Background] Tanaka Y, Matsumoto I, Iwanami K, Inoue A, Umeda N, Tanaka Y, Sugihara M, Hayashi T, Ito S, Sumida T. Six-transmembrane epithelial antigen of prostate 4 (STEAP4) is expressed on monocytes/neutrophils, and is regulated by TNF antagonist in patients with rheumatoid arthritis. Clin Exp Rheumatol. 2012 Jan-Feb;30(1):99-102. Epub 2012 Mar 6. PMID 22244520
- [Background] Daien CI, Morel J. Predictive factors of response to biological disease modifying antirheumatic drugs: towards personalized medicine. Mediators Inflamm. 2014;2014:386148. doi: 10.1155/2014/386148. Epub 2014 Jan 12. PMID 24523570
- [Background] Kristensen LE, Bliddal H, Christensen R, Karlsson JA, Gulfe A, Saxne T, Geborek P. Is swollen to tender joint count ratio a new and useful clinical marker for biologic drug response in rheumatoid arthritis? Results from a Swedish cohort. Arthritis Care Res (Hoboken). 2014 Feb;66(2):173-9. doi: 10.1002/acr.22107. PMID 23982986
- [Background] Xie X, Zhang D, Chen JW, Tian J, Ling GH, Li F. Pharmacogenomics of biological treatment in rheumatoid arthritis. Expert Opin Biol Ther. 2014 Feb;14(2):157-64. doi: 10.1517/14712598.2014.859672. Epub 2013 Dec 3. PMID 24295560